CLINICAL TRIAL: NCT00122993
Title: Worksite Environmental Interventions for Weight Control
Brief Title: Worksite Program to Prevent Weight Gain Among Bus Drivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 0409S63606; R01HL079478 (NIH)
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Obesity; Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Obesity; Cardiovascular Diseases; Heart Diseases | interventions — Commerce; Exercise; Environment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Multi-component environmental intervention to prevent excess weight gain among bus drivers
  Interventions: Behavioral: Healthful eating and food choices behavior change programs and changes in worksite food availability and prices; Behavioral: Physical Activity; Behavioral: Environment
- 2 (No Intervention): Control group

INTERVENTIONS:
Behavioral: Healthful eating and food choices behavior change programs and changes in worksite food availability and prices — Food choices and eating behavior programs and environmental changes will be implemented for 18 months in intervention garages.
  Arms: 1
Behavioral: Physical Activity — Physical activity programs are offered at the intervention garages for an 18 month period.
  Arms: 1
Behavioral: Environment — Changes in the food and physical activity environment are made for an 18 month period in intervention garages. These include improving the healthfulness of the foods available in vending machines, and improving the fitness rooms at the garages.
  Arms: 1

SUMMARY:
The purpose of this study is to implement and evaluate a two-year multi-component environmental intervention to prevent weight gain among city bus drivers at four bus garages.

It is hypothesized that transit employees in the intervention garages will gain less weight compared to the transit employees in the control garages.

DETAILED DESCRIPTION:
BACKGROUND:

Environmental influences that support less healthful food choices and sedentary behaviors have contributed to the epidemic increase in overweight and obesity among U.S. adults. Worksite settings are an effective channel through which to reach adults with interventions designed to prevent excess weight gain and obesity.

DESIGN NARRATIVE:

This study will implement and evaluate a multi-component environmental intervention to prevent excess weight gain among 1200 bus drivers working in four garages in a major metropolitan area. Four garages will be randomized to the intervention or control group for a two-year period. The environmental interventions are based on a social ecological framework and target four worksite environmental areas: 1) food availability and incentives; 2) physical activity opportunities and incentives; 3) the social environment; and 4) media/promotion related to health food choices, physical activity, and body weight.

ELIGIBILITY:
Inclusion Criteria:

* Employed as a bus driver

Exclusion criteria:

* Not employed as a bus operator at one of the four participating garages

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2004-09; Primary Completion 2007-12 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Change in body weight | Measured at Year 2

SECONDARY OUTCOMES:
Changes in energy intake and physical activity | Measured at Year 2
Health claims cost | Measured at Year 2

CONTACTS AND LOCATIONS:
Overall Officials: Simone French, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States